CLINICAL TRIAL: NCT03118037
Title: Transcervical Radiofrequency Ablation of Uterine Fibroids Global Registry (SAGE)
Brief Title: Transcervical Radiofrequency Ablation of Uterine Fibroids Global Registry
Acronym: SAGE
Status: Terminated | Type: Observational
Why Stopped: Termination due to continued lack of patient compliance
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Other Study IDs: CL 04878
Record Dates: First submitted 2017-03-27; First posted 2017-04-18 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Uterine Fibroid
Keywords: Radiofrequency Ablation
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Sonata: Women who undergo transcervical radiofrequency(RF) ablation with the Sonata System for treatment of their fibroids
  Interventions: Device: Sonata System

INTERVENTIONS:
Device: Sonata System — Transcervical access for radiofrequency ablation of uterine fibroids
  Other Names: Transcervical RF Ablation

SUMMARY:
SAGE is an observational post market registry with the objective of characterizing long term outcomes after treatment of uterine fibroids with the Sonata System in real world clinical practice settings.

DETAILED DESCRIPTION:
Patients whom have selected the CE-marked Sonata system for treatment of fibroids will be approached for study participation. Participation in the trial will consist of data collection in the form of questionnaires prior to and after the treatment at the following intervals: pre-procedure, 4 weeks, 1, 2, 3, 4 and 5 years following treatment.

The following data points will be collected: Length of stay, time to return to normal activities (Treatment Recovery Questionnaire), time to return to sexual activity (Treatment Recovery Questionnaire), change in fibroid symptom severity and quality of life (UFS-QOL), change in general health outcome (EQ-5D), work productivity and activity impairment (WPAI), subject satisfaction and overall treatment effect (Overall Treatment Effect and Satisfaction Questionnaire), pregnancy occurrence and outcome, non-medical re-intervention, adverse events related to the device/procedure.

Validated questionnaires are used where appropriate (UFS-QOL, E1-5D and WPAI). Double data entry will occur to ensure accurate capture of subject reported data. Monitoring will occur throughout the course of the trial to ensure adherence to the protocol.

As an observational trial, there are no pre-specified statistically powered endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Have selected Sonata for treatment of symptomatic uterine fibroids or is participating in the OPEN study (Evaluation of Uterine Patency Following Sonography-guided Transcervical Ablation of Fibroids, NCT02844920, protocol # CL04897) or has completed participation in the OPEN study within the last 14 months
* Speaks and reads a language for which questionnaires are available
* Are greater than or equal to 18 years of age at the time of enrollment
* Willing and able to read, understand and sign the informed consent form, to participate in the registry and to adhere to all registry study follow-up requirements

Exclusion Criteria:

* Any reason for which, in the opinion of the Investigator, the individual study patient is not appropriate or suitable for participation in the registry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women with diagnosed uterine fibroids are eligible to participate
Study Population: Women who select to have their uterine fibroids treated with the Sonata System
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Pregnancy and Pregnancy Outcomes | Up to 5 years-post procedure
  Number of subjects with pregnancy and the number of pregnancies during the 5 year follow-up period. Outcome of each pregnancy including pregnancy outcomes, delivery route, antenatal and perinatal complications.
Surgical Re-intervention for Heavy Menstrual Bleeding | Up to 5 years-post procedure
  Number of subjects who had surgical re-intervention to treat heavy menstrual bleeding during the 5 year follow-up period.

OTHER OUTCOMES:
Uterine Fibroid Symptom - Quality of Life | Pre-procedure and up to 5 years
  UFS-QoL, validated fibroid specific assessment tool
Length of Stay | From admission to hospital discharge, up to four weeks.
  Length of stay (in hours) for the treatment of fibroids with the Sonata System (which occurs at enrollment into the registry).
Time to Return to Normal Daily Activity | First two weeks post procedure
  Questionnaire
Time to Return to Sexual Activity | First two weeks post procedure
  Questionnaire
Change in General Health Outcome | Pre-procedure and up to 5 years
  EQ-5D standardized instrument for use as a measure of health outcome
Work Productivity and Activity Impairment | Pre-procedure and up to 5 years
  Standardized instrument for assessing activity/productivity impairment, commonly used in health economics outcomes research. The tool measure impairment in percentage.
Subject Satisfaction | At 1 year post procedure and up to 5 years
  Questionnaire
Overall Treatment Effect | At 1 year post procedure and up to 5 years
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (6):
  - Evangelisches Krankenhaus Köln-Weyertal gemeinnützige GmbH, Cologne
  - Frauenklinik Universitätsklinikum Jena, Jena
  - Klinik für Frauenheilkunde und Geburtshilfe, Kempten
  - MarienKrankenhaus Schwerte Frauenklinik, Schwerte
  - Josephs-Hospital Warendorf, Warendorf
  - Marien Hospital Witten, Witten
- Spital Oberengadin, Samedan, Switzerland
- United Kingdom (2):
  - Addenbrookes Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Liverpool Women's NHS Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christoffel L, Romer T, Schiermeier S. Transcervical Radiofrequency Ablation of Uterine Fibroids Global Registry (SAGE): Study Protocol and Preliminary Results. Med Devices (Auckl). 2021 Mar 3;14:77-84. doi: 10.2147/MDER.S301166. eCollection 2021. PMID 33688276